CLINICAL TRIAL: NCT04001439
Title: FEcal Microbiota Transplantation for MAjor Depression in Schizophrenia (FEMADSZ)
Brief Title: FEcal Microbiota Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-11; 2019-11 (Registry Identifier: APHM)
Record Dates: First submitted 2019-06-20; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Depression in Schizophrenia
MeSH Terms: interventions — Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: All patients will receive 30 microbiota capsules in take proceded by bowel lavage by 4 liters macrogo solution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical trial (Other): the study design is an open-label, single-arm propective clinical trial. In this proof-of-concept study we will assess feasibility safety and potential efficacy of an intervention of FMT in SZ subjects with MD.
  Interventions: Drug: Experimental drug

INTERVENTIONS:
Drug: Experimental drug — All patients will recive 30 microbiota capsules intake preceded by bowel lavage by 4 liters macrogol solution. the capsules are developed by the services of JC Lagier.

SUMMARY:
The primary objective will be to evaluate effectiveness, safety and acceptability of FMT on depressive symptoms at 2 months follow-up in SZ patients with resistant MD.

DETAILED DESCRIPTION:
Background. Major Depression (MD) will move into the first place of cause of the global burden of disease by 2030. Conventional treatments (antidepressants) are only partly effective with frequent side effects. More specifically, MD is underdiagnosed and undertreated in schizophrenia (SZ) despite its high impact on prognosis and quality of life in SZ patients. Even when treated, 44% of the patients remain major depressed under conventional antidepressants.

FEMADSZ makes the hypothesis that this is due to the fact that the source of MD relies outside the brain, in the gut microbiota. The associations between microbiota disturbances are now well demonstrated in rodent models (>60 studies) and indirect data in humans clearly suggest that the microbiota hypothesis of MD is the most promising track in psychiatry. The primary objective will be to evaluate effectiveness, safety and acceptability of FMT on depressive symptoms at 2 months follow-up in SZ patients with resistant MD. Methods: This is a pilot, single-arm, prospective, open-label proof-of-concept trial, including SZ patients with resistant MD. Fifteen patients will be enrolled and administered a Fecal Microbiota Transplantation. The main outcome measure will be depressive score at 2 months, adverse events and acceptability. Each patient will receive a FDG-PET scan, a routine blood draw and a metagenomic microbiota analysis before and after intervention. Expected results. This pilot study will help determining the effectiveness of FMT and the neurobiologic and microbiologic mechanisms associated with response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 65 years
* with the current diagnosis of shizophrenia

Exclusion Criteria:

* history of lifetime FMT
* History of gut surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3088 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
myoglobin concentration | 2 moths
  the primary outcome for efficacy will be the improvement of depressive symtoms